CLINICAL TRIAL: NCT01773226
Title: A Prospective Single-Center Clinical Study of a Single Intra-Articular Injection of Autologous Protein Solution ("APS(TM)") in Patients With Osteoarthritis (OA) of the Knee
Brief Title: Evaluation of Intra-articular Injection of Autologous Protein Solution ("APS(TM)") for the Treatment of Osteoarthritis (OA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APSS-11-00
Record Dates: First submitted 2013-01-07; First posted 2013-01-23 (Estimated); Results first posted 2016-06-15 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Gonarthrosis; Knee Osteoarthritis; Osteoarthritis
Keywords: Autologous Protein Solution; APS; Osteoarthritis; Injection
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous Protein Solution "APS(TM)" (Experimental): Patients who have been treated with a single, intra-articular injection.
  Interventions: Device: Autologous Protein Solution "APS(TM)"

INTERVENTIONS:
Device: Autologous Protein Solution "APS(TM)" — A therapy prepared at the point-of-care from a small sample of the patient's own blood containing high concentrations of anti-inflammatory and anabolic proteins

SUMMARY:
This prospective single-center study will evaluate the safety and tolerability of a single dose of "APS(TM)" treated patients with OA of the knee who have failed conservative OA therapy. The study will also evaluate efficacy by assessing patient pain and functionality.

ELIGIBILITY:
Eligibility Criteria:

* Male or female ≥40 years.
* Willingness and ability to comply with the study procedures and visit schedules and ability to follow verbal and written instructions.
* A standing radiograph of the knee showing a Kellgren grade of 2 or 3
* Frequency of knee pain on most days over the last month.
* Diagnosis of unilateral knee OA
* Body mass index (BMI) ≤40 kg/m2.
* Failed conservative OA therapy.
* Signed an independent ethics committee (IEC)-approved informed consent form (ICF).
* Willingness to abstain from the use of topical pain therapies, intra-articular corticosteroids, and viscosupplementation during the study.
* Willingness to abstain from systemic pain medications except rescue medication.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R.A.M. van Drumpt, M.D., Principal Investigator — St. Anna Hospital, Geldrop, NL
Locations (1):
- St. Anna Hospital, Geldrop, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] King W, van der Weegen W, Van Drumpt R, Soons H, Toler K, Woodell-May J. White blood cell concentration correlates with increased concentrations of IL-1ra and improvement in WOMAC pain scores in an open-label safety study of autologous protein solution. J Exp Orthop. 2016 Dec;3(1):9. doi: 10.1186/s40634-016-0043-7. Epub 2016 Feb 9. PMID 26915009

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single-centre study in the Netherlands. FPI April 2013.
Pre-assignment Details: All patients treated with APS who had at least 1 post-injection assessment of clinical outcomes were to be included in the clinical outcomes population, which was used for the clinical outcomes summaries and listings
Period: Overall Study
Arm/Group | Autologous Protein Solution "APS(TM)"
Started | 11
Completed | 10 (Withdrawal of one subject after one-month assessment due to persistent OA symptoms)
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Autologous Protein Solution "APS(TM)"
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Region of Enrollment [Number; unit: participants]
  Netherlands | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: Safety and tolerability will be assessed from AEs and injection-site reactions, physical examinations, knee examinations, vital signs, ECGs, and clinical laboratory tests (hematology, coagulation, blood chemistry, and urinalysis) evaluated at baseline (pre-injection) and post-injection up to 6 months.
Time Frame: Up to 6 months post-injection
Population: In cases where a patient reported multiple occurrences of an AE, the first occurrence of the worst reported case of the event was to be used for the purpose of analysis.
Measure: Number; unit: Adverse Events (AEs)
Arm/Group | Autologous Protein Solution "APS(TM)"
Number analyzed (Participants) | 11
Adverse Events (AEs) | 22

2. Secondary Outcome: Number of Patients Using Rescue Medication
Description: Explore the potential for an analgesic effect of a single dose of APS in patients with OA of the knee.
Time Frame: Up to 6 months post-injection
Population: The incidence of patients using rescue medication for OA pain.
Measure: Number; unit: Frequency of Patients using Rescue medic
Arm/Group | Autologous Protein Solution "APS(TM)"
Number analyzed (Participants) | 11
Frequency of Patients using Rescue medic
  Injection visit | 2
  Month 6 | 2

3. Secondary Outcome: Pain Score
Description: The Western Ontario and McMaster Universities osteoarthritis index questionnaire using the Likert scale (WOMAC LK), Version 3.1 questionnaire has 24 items that the patient addresses about the knee: 5 items on the pain subscale, 2 on the stiffness subscale, and 17 on the physical function subscale. Each item was to be answered on a 5-point Likert scale, with grading from 0 (none or never) to 4 (extreme or always). The scores are summed for items in each subscale, with possible ranges as follows: pain=0-20, stiffness=0-8, physical function=0-68. A higher score indicates worse pain, stiffness, or functional limitation.
Time Frame: Baseline, Week 1, Week 2, and at Months 1, 3, and 6.
Population: Results of the WOMAC LK 3.1 questionnaire (pain, stiffness, and functionality subscores) were summarized by timepoint.
Measure: Mean (Standard Deviation); unit: Scores on a WOMAC pain scale
Arm/Group | Autologous Protein Solution "APS(TM)"
Number analyzed (Participants) | 11
Scores on a WOMAC pain scale
  Baseline | 12 (1.6)
  Week 1 | 8.2 (5.1)
  Week 2 | 6.5 (4.7)
  Month 1 | 4.5 (4.1)
  Month 3 | 3.0 (3.1)
  Month 6 | 3.1 (4.3)

4. Secondary Outcome: Stiffness Score
Description: Changed Outcome Measure Description to: The Western Ontario and McMaster Universities osteoarthritis index questionnaire using the Likert scale (WOMAC LK), Version 3.1 questionnaire has 24 items that the patient addresses about the knee: 5 items on the pain subscale, 2 on the stiffness subscale, and 17 on the physical function subscale. Each item was to be answered on a 5-point Likert scale, with grading from 0 (none or never) to 4 (extreme or always). The scores are summed for items in each subscale, with possible ranges as follows: pain=0-20, stiffness=0-8, physical function=0-68. A higher score indicates worse pain, stiffness, or functional limitation.
Time Frame: Baseline, Week 1, Week 2, and at Months 1, 3, and 6.
Population: Results of the WOMAC LK 3.1 questionnaire (pain, stiffness, and functionality subscores) were summarized by timepoint.
Measure: Mean (Standard Deviation); unit: Scores on a WOMAC stiffness scale
Arm/Group | Autologous Protein Solution "APS(TM)"
Number analyzed (Participants) | 11
Scores on a WOMAC stiffness scale
  Baseline | 4.9 (0.9)
  Week 1 | 3.8 (1.7)
  Week 2 | 3.1 (1.2)
  Month 1 | 2.5 (1.8)
  Month 3 | 1.7 (1.8)
  Month 6 | 2.3 (1.9)

5. Secondary Outcome: Physical Function Score
Description: as for outcome 4
Time Frame: Baseline, Week 1, Week 2, and at Months 1, 3, and 6.
Population: Results of the WOMAC LK 3.1 questionnaire (pain, stiffness, and functionality subscores) were summarized by timepoint.
Measure: Mean (Standard Deviation); unit: Scores on a WOMAC functionality scale
Arm/Group | Autologous Protein Solution "APS(TM)"
Number analyzed (Participants) | 11
Scores on a WOMAC functionality scale
  Baseline | 38.1 (7.5)
  Week 1 | 27.8 (16.2)
  Week 2 | 21.9 (13.4)
  Month 1 | 17.5 (15.1)
  Month 3 | 10 (11.4)
  Month 6 | 12.3 (14.7)

ADVERSE EVENTS:
Time Frame: AEs were recorded at each visit (Week 1, Week 2, Month 1, Month 3, Month 6)
Description: In cases where a patient reported multiple occurrences of an AE, the first occurrence of the worst reported case of the event was to be used for the purpose of analysis.
Arm/Group | Autologous Protein Solution "APS(TM)"
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 9/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Protein Solution "APS(TM)" (N=11)
Joint effusion (Musculoskeletal and connective tissue disorders) | 6 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 3 (3)
Joint instability (Musculoskeletal and connective tissue disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Site Discomfort (General disorders) | 1 (1)
Injection site joint pain (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Tootache (Gastrointestinal disorders) | 1 (1)
Procedural Nausea (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
1. Small sample size
2. Unblinded observational study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less